CLINICAL TRIAL: NCT06468826
Title: A Phase 1, Open-label, Single-dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Avacopan in Subjects With Normal Renal Function and Subjects With End-Stage Renal Disease (ESRD) Requiring Hemodialysis
Brief Title: A Study of Avacopan in Participants With Normal Renal Function and Participants With End-Stage Renal Disease (ESRD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20230265
Record Dates: First submitted 2024-06-17; First posted 2024-06-21 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: End-Stage Renal Disease (ESRD)
Keywords: End-Stage Renal Disease; ESRD; Renal Function; Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — avacopan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Normal Renal Function (Experimental): Participants in Group 1 will receive a single dose of avacopan on Day 1.
  Interventions: Drug: Avacopan
- Group 2: ESRD Requiring HD (Experimental): Participants in Group 2 will receive a single dose of avacopan on Day 1 in each of 2 treatment periods (Period 1/on HD and Period 2/off HD).
  Interventions: Drug: Avacopan

INTERVENTIONS:
Drug: Avacopan — Oral capsules
  Other Names: Tavneos; AMG 569; CCX168

SUMMARY:
The primary objective of the study is to evaluate the pharmacokinetics (PK) of avacopan and metabolite (M1) after a single dose of avacopan in participants with normal renal function and participants with ESRD requiring hemodialysis (HD).

ELIGIBILITY:
Inclusion Criteria

* Participant has provided informed consent.
* Male or female participants, between 18 and 75 years of age (inclusive) at the time of Screening.
* Body mass index between 18 and <40 kg/m^2 at the time of Screening.
* Eligible participants will be classified based on established need for renal replacement therapy and estimated glomerular filtration rate (eGFR).

  1. Group 1 (normal renal function): eGFR ≥90 mL/min and no history of renal disease.
  2. Group 2 (ESRD requiring HD): eGFR <15 mL/min and receiving HD.

Exclusion Criteria

All Participants:

* History of uncontrolled or unstable cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, hematopoietic, psychiatric, or neurological disease, or evidence of rapidly deteriorating renal function.
* History or evidence, at Screening or Check-in, of clinically significant disorder, condition, or disease not otherwise excluded that, in the opinion of the Investigator (or designee), would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion.
* Total white blood cell count is below the lower limit of normal at Screening or Check-in.
* Significant infection within 28 days before Check-in.
* Prior infection with or exposure to tuberculosis, or travel to areas of endemic tuberculosis or endemic mycoses within the past 6 months.
* Active liver disease or hepatic dysfunction, defined as aspartate aminotransferase or alanine aminotransferase > the upper limit of normal for Group 1 (normal renal function) and >2 times the upper limit of normal for Group 2 (ESRD requiring HD).
* History or evidence, at Screening or Check-in, of poorly controlled diabetes (regardless of type), based on hemoglobin A1C of >10%.
* Clinically significant hyperkalemia (defined by serum potassium concentration as >5.5 mEq/L for Group 1 [normal renal function], >6 mEq/L for Group 2 [ESRD requiring HD]) at Screening or Check-in.
* Participants who have a current, functioning organ transplant and/or are on immunosuppressants.
* Participants on the national transplant list (United Network for Organ Sharing) at Screening who anticipate receiving an organ transplant within 4 months.
* Positive human immunodeficiency virus test.
* Positive hepatitis B or hepatitis C panel at Screening. Participants whose results are compatible with prior hepatitis B infection (positive hepatitis B surface antibody, positive hepatitis B core antibody, or negative HBsAg) will be excluded. Participants whose results are compatible with prior hepatitis B vaccination may be included.
* History or evidence of clinically significant arrhythmia at Screening, including any clinically significant findings on the ECG taken at Check-in.
* History suggestive of esophageal (including esophageal spasm, esophagitis), gastric, or duodenal ulceration, or bowel disease (including but not limited to peptic ulceration, gastrointestinal bleeding, ulcerative colitis, Crohn's disease, or irritable bowel syndrome); or a history of gastrointestinal surgery, other than uncomplicated appendectomy.
* Female participants with a positive pregnancy test at Screening or Check-in.
* Female participants lactating/breastfeeding or who plan to breastfeed during the study through 60 days after administration of investigational product.

Participants in Group 1 (normal renal function) are excluded if:

* History of malignancy of any type, with the exception of the following: in situ cervical cancer or surgically excised non-melanomatous skin cancers more than 5 years before receiving avacopan.
* A corrected QT interval by Fredericia (QTcF) >450 msec in males or >470 msec in females or history/evidence of long QT syndrome at Screening or Check-in.
* A history of renal disease or renal injury as indicated by medical history or an abnormal renal function profile at Screening or Check-in.

Participants in Group 2 (ESRD requiring HD) are excluded if:

* Child-Pugh classification of Class C. Child-Pugh will only be evaluated for participants deemed to have active liver disease by the Investigator (or designee).
* Active malignancy of any type.
* A change in disease status within 30 days of Screening, as documented by the participants medical history, deemed clinically significant by the Investigator.
* A QTcF ≥470 msec in males or ≥480 msec in females.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2024-07-11 (Actual); Primary Completion 2024-10-05 (Actual); Study Completion 2024-10-05 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Avacopan | Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36 hours (postdose), Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 12, Day 15, and Day 18.
Cmax of M1 | Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36 hours (postdose), Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 12, Day 15, and Day 18.
Area Under the Plasma Concentration-time Curve (AUC) from Time Zero to Time of Last Quantifiable Concentration (AUClast) of Avacopan | Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36 hours (postdose), Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 12, Day 15, and Day 18.
AUClast of M1 | Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36 hours (postdose), Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 12, Day 15, and Day 18.
AUC from Time Zero to Infinity (AUCinf) of Avacopan | Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36 hours (postdose), Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 12, Day 15, and Day 18.
AUCinf of M1 | Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36 hours (postdose), Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 12, Day 15, and Day 18.
AUC from Time Zero to 48 Hours (AUC0-48) of Avacopan | Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36 hours (postdose), Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 12, Day 15, and Day 18.
AUC0-48 of M1 | Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36 hours (postdose), Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 12, Day 15, and Day 18.
HD Clearance of Drug Dialysate (CLD) of Avacopan | Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36 hours (postdose), Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 12, Day 15, and Day 18.
HD CLD of M1 | Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36 hours (postdose), Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 12, Day 15, and Day 18.

SECONDARY OUTCOMES:
Number of Participants who Experienced Treatment-emergent Adverse Events | Up to approximately 37 days.
Number of Participants who Experienced Serious Adverse Events | Up to approximately 96 days.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (2):
- United States (2):
  - Floridian Clinical Research, LLC, Miami Lakes, Florida
  - Orlando Clinical Research Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com